CLINICAL TRIAL: NCT03282435
Title: Treatment of Non-small Cell Lung Cancer With CIK Cells Blocked by PD-1 Antibody
Brief Title: Treatment of Non-small Cell Lung Cancer With Cytokine-induced Killer (CIK) Cells Blocked by PD-1 Antibody
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dalian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: zsyy_zxsys2018-01
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIK cells with PD-1 blocking (Experimental): CIK cellular therapy with PD-1 blocking combined with standard lung cancer treatment
  Interventions: Biological: CIK cells with PD-1 blocking; Other: standard lung cancer treament
- CIK cells without PD-1 blocking (Active Comparator): CIK cellular therapy without PD-1 blocking combined with the same standard lung cancer treatment as the experimental group patients receive
  Interventions: Other: standard lung cancer treament; Biological: CIK cells without PD-1 blocking

INTERVENTIONS:
Biological: CIK cells with PD-1 blocking — CIK cellular therapy with PD-1 blocking
  Arms: CIK cells with PD-1 blocking
Other: standard lung cancer treament — standard non-small cell lung cancer treatment: surgery, chemotherapy
Biological: CIK cells without PD-1 blocking — CIK cellular therapy without PD-1 blocking
  Arms: CIK cells without PD-1 blocking

SUMMARY:
to evaluate the prognosis of non-small cell lung carcinoma patients under CIK cellular treatment with PD-1 blocking on top of the standard therapy

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer;
* more than 50% tumor tissues positive with PD-L1;
* EGFR and ALK wild type
* no other tumors

Exclusion Criteria:

* with systematic diseases shortening survival

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5 years
metastasis-free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: xiaolin Yuan, Principal Investigator — Affiliated Zhongshan Hospital of Dalian University

IPD SHARING:
Plan to Share IPD: Yes
age, gender, tumor staging